CLINICAL TRIAL: NCT05683509
Title: Biologically Oriented Alveolar Ridge Preservation With Layered Collagen and Xenograft (A Randomized Controlled Clinical Trial With Histological Evaluation)
Brief Title: Alveolar Ridge Preservation With Layered Collagen and Xenograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD-992
Record Dates: First submitted 2022-12-12; First posted 2023-01-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-01

CONDITIONS: Alveolar Ridge Preservation
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: The application of deep collagen layer, xenograft and collagen membrane seal versus the use of xenograft and collagen membrane seal alone in alveolar ridge preservation procedures.
Who Masked: Outcomes Assessor
Masking Description: the outcome assessor will be blinded about the grouping and which patient got which treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- deep collagen layer, xenograft and collagen membrane (Active Comparator): Alveolar ridge preservation is done using deep collagen layer, xenograft and collagen membrane
  Interventions: Procedure: deep collagen layer, xenograft and collagen membrane
- xenograft and collagen membrane (Active Comparator): Alveolar ridge preservation is done using xenograft and collagen membrane alone
  Interventions: Procedure: xenograft and collagen membrane

INTERVENTIONS:
Procedure: deep collagen layer, xenograft and collagen membrane — Alveolar ridge preservation is done using deep collagen layer, xenograft and collagen membrane
  Arms: deep collagen layer, xenograft and collagen membrane
Procedure: xenograft and collagen membrane — Alveolar ridge preservation is done using xenograft and collagen membrane only
  Arms: xenograft and collagen membrane

SUMMARY:
alveolar ridge preservation using deep collagen layer, xenograft and collagen membrane seal versus the use of xenograft and collagen membrane seal alone. Measuring the clinical and radiographic alveolar ridge dimensional changes following after preservation at the time of implant placement

DETAILED DESCRIPTION:
alveolar ridge preservation using deep collagen layer, xenograft and collagen membrane seal versus the use of xenograft and collagen membrane seal alone.

The primary objective of the study is measuring the clinical and radiographic alveolar ridge dimensional changes following the procedure 4 months post operatively

The secondary objective :

* Histological assessment of alveolar bone specimens to assess bone remodeling and new bone formation in both studied groups after four months.
* Patient satisfaction after implant placement

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (American Society of Anesthesiologists I; ASA I).

  * Patients diagnosed with single unrestorable molar teeth (socket type I) requiring extraction and implant placement (Elian et al.2007).
* Teeth free from any infection or periapical pathosis.
* Enough zone of keratinized tissue with at least 2mm.
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow up and maintenance program.

Exclusion Criteria:

* Bad oral hygiene.
* Presence of smoking habit.
* Presence of occlusal interferences
* Pregnant females
* Vulnerable group of patients (handicapped, mentally retarded and prisoners) (according to the recommendation of esthetical committee of Faculty of Dentistry Ain Shams University).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Measuring the clinical alveolar ridge changes | at baseline and 4 months
  Measuring the thickness of the alveolar ridge in mm
Measuring the radiographic change in the buccal bone thickness | at baseline and 4 months
  Measuring the change in the thickness of the buccal ridge radiographically in mm
Measuring the radiographic alveolar ridge dimensional changes | at baseline and 4 months
  Measuring the bone density in hounsfield units (HU)

SECONDARY OUTCOMES:
Histological assessment of core biopsy | 4 months post operatively
  The microscopic examination of the bone remodeling and new bone through tissue biopsy (fixation and staining of the tissues) to examine the newly formed cells and count them to determine the amount of newly tissue formed

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abu el ela, Prof, Study Chair — Faculty of dentistry ain shams university
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No